CLINICAL TRIAL: NCT01725737
Title: Placebo-Controlled Trial With GlyTI-M Among Children With ADHD
Brief Title: Placebo-Controlled Trial With GlyTI-M Among Children With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ruu-Fen Tzang, attending physician, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09MMHIS178; 09MMHIS178 (Other: 09MMHIS178)
Record Dates: First submitted 2012-11-06; First posted 2012-11-14 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: ADHD
Keywords: ADHD; GlyTI-M
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- GlyTI-M (Active Comparator): GlyTI-M: 0.03gm/kg/day
  Interventions: Drug: GlyTI-M

INTERVENTIONS:
Drug: GlyTI-M
  Arms: GlyTI-M
Drug: Placebo — Placebo Comparator: starch
  Arms: Placebo

SUMMARY:
Although psychostimulant is the first line of drug to treat Attention Deficit Hyperactivity Disorder, (ADHD), actually there are 10-20% ADHD patient do not response well to current medication. Most of parents of children with ADHD in Taiwan dislike to use psychostimulant. We expect that GlyTI-M will have better efficacy than placebo to reduce ADHD symptoms. This study will also help us to understand the mechanism of ADHD and give a way to develop new drug and also a more possible way to treat ADHD children under 6 years old.

DETAILED DESCRIPTION:
The accumulated neuro-image, hereditary and animal studies showed the correlation between glutamate transport dysfunction and ADHD psychopathology. However, there is limited clinical trial to testify the effect of modulating the NMDA receptor function of glutamate to treat ADHD.

GlyTI-M is an endogenous Glycine transporter I inhibitor, and it acts on the glutamatergic synapse to modulate the neurotransmission of N-Methyl-D-Aspertate (NMDA) receptor. This study aims to explore the effect of GlyTI-M among children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the criteria of ADHD according to the Diagnostic and Statistic Manual, fourth edition (DSM-IV).
* Subjects and parents agree to participate in the study and provide informed consent.

Exclusion Criteria:

* Autism, Mental retardation.
* inability to follow protocol.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2012-04; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Swanson, Nolan, and Pelham, version IV scale (SNAP-IV-C) | 1. Change from Baseline in inattention, hyperactivity/impulsivity , oppositional defiant disorder score of SNAP-IV-C at 0, 2, 4, 6week
  1. Change in inattention score of SNAP-IV-C
  2. Change in hyperactivity/impulsivity score of SNAP-IV-C
  3. Change in oppositional defiant disorder score of SNAP-IV-C

SECONDARY OUTCOMES:
Barkley's side effect rating scale | 1. Change from Baseline adverse effect at 2, 4, 6 weeks
  1. Change from Baseline adverse effect at 2 weeks
  2. Change from Baseline adverse effect at 4 weeks
  3. Change from Baseline adverse effect at 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ruu-Fen Tzang, M.D., Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taipei, Taiwan